CLINICAL TRIAL: NCT06226129
Title: Gadopiclenol (Elucirem): A New Gadolinium Based Contrast Agent With High Relaxivity for Increased Contrast and Improved Differentiation of Clinically Significant Prostate Cancer on Contrast Enhanced MRI: A Prospective Study.
Brief Title: Gadopiclenol in Contrast Enhanced MRI of the Prostate
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Guerbet (Industry)
Responsible Party: Principal Investigator, Nicolas Bloch, Professor of Radiology, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAV5623
Record Dates: First submitted 2024-01-02; First posted 2024-01-26 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer
Keywords: MRI; Prostate; Contrast Agent
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gadopiclenol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gadopiclenol (Experimental): Gadopiclenol in dose, route of administration, and indication that is FDA-approved.
  Interventions: Drug: Gadopiclenol

INTERVENTIONS:
Drug: Gadopiclenol — Gadopiclenol for contrast enhanced MRI

SUMMARY:
The fundamental aim of this study is to show that the novel contrast agent Gadopiclenol (Elucirem), with its high relaxivity, facilitates increased contrast enhancement and improved differentiation of clinically significant prostate cancer on Prostate MRI, as categorized by the PI-RADS v2 classification categories.

DETAILED DESCRIPTION:
Gadolinium based contrast agents with higher relaxivity have been shown to improve contrast enhancement and differentiation of tissues with increased blood perfusion or with higher microvascular density (MVD), and therefore increase visibility of cancerous tissue. In this study, the objective is to demonstrate that Gadopiclenol facilitates the detection and classification of clinically significant prostate cancer, compared to T2-W (T2 weighted image) and diffusion weighted imaging (DWI), using the detailed location-specific (individual biopsy core for each annotated target) results of subsequently performed MRI-US fusion biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo a clinically indicated MRI of the prostate with contrast.
* Scheduled to undergo, or likely to be scheduled to undergo, a prostate MRI-US fusion biopsy with histology results available within 6 months of their MRI.

Exclusion Criteria:

* Prisoner
* Have already begun therapeutic treatment for prostate cancer including surgery (TURP, prostatectomy), radiotherapy, hormone therapy or chemotherapy.
* Patients with end stage renal failure who are on dialysis. Patients who have chronic kidney disease or acute kidney injury are contraindicated for MRI per FDA and ACR (American College of Radiologists) guidelines and would thus be excluded as well.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Blinded Radiology Review of Enhancement of Images, Graded 1-5 | Through Study Completion (An Average of 1 Year Post-MRI)
  Single qualitative grade for contrast enhancement quality, with each exam being graded on a scale of 1-(Fail) to 5-(Excellent) contrast enhancement quality.

SECONDARY OUTCOMES:
Quantitative Measurements of Wash-In/Wash-Out Contrast Curve | Through Study Completion (An Average of 1 Year Post-MRI)
  The secondary outcomes will be the quantitative measurement of the wash-in/wash-out contrast curve of the individual PI-RADS lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Bloch, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No